CLINICAL TRIAL: NCT05453136
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled Phase 3 Study of TS-142 in Patients with Insomnia Disorder.
Brief Title: Phase III Study of TS-142 in Patients with Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS142-301
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-09

CONDITIONS: Patients with Insomnia
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5 mg (Experimental): Period in which participants received repeated doses of 5 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142 5 mg
- 10 mg (Experimental): Period in which participants received repeated doses of 10 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142 10 mg
- Placebo (Placebo Comparator): Period in which participants received repeated doses of placebo prior to bedtime
  Interventions: Drug: Placebo to TS-142

INTERVENTIONS:
Drug: TS-142 5 mg — Participants received repeated doses of 5 mg of TS-142 (oral tablet)
  Arms: 5 mg
Drug: TS-142 10 mg — Participants received repeated doses of 10 mg of TS-142 (oral tablet)
  Arms: 10 mg
Drug: Placebo to TS-142 — Participants received repeated doses of placebo to TS-142 (oral tablet)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multi-center, placebo-controlled, parallel-group confirmatory study in patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male and female who are aged 18 years or older at the time of informed consent
2. Outpatients
3. Patients falling under the category of insomnia disorder according to the diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)

Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. Patients falling under the category of any disorders other than insomnia disorder among sleep-wake disorders according to the diagnostic criteria in DSM-5
2. Patients with psychiatric disorders such as depression, schizophrenia, and anxiety
3. Patients with difficulty sleeping due to medical problems such as pain, pruritus, hot flush, nocturia (> 3 times per night), heart disease, bronchial asthma, reflux esophagitis, endocrine disease, and periodic limb movement disorder

Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1155 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Difference of subjective sleep latency (sSL) between TS-142 and placebo in mean change from baseline | Baseline and Week 2
  sSL is defined as the duration of time until which subjects fall asleep recorded in a sleep diary.

SECONDARY OUTCOMES:
Difference of subjective sleep efficacy (sSE) between TS-142 and placebo in mean change from baseline | Baseline and Week 2
  sSE is defined as the percentage of subjective total sleep time (sTST) in total amount of time from bedtime to wake-up time in a sleep diary.
Difference of sTST between TS-142 and placebo in mean change from baseline | Baseline and Week 2
  sTST is defined as the total amount of time spent asleep before wake-up time as recorded in a sleep diary.
Difference of subjective wake time after sleep onset (sWASO) between TS-142 and placebo in mean change from baseline | Baseline and Week 2
  sWASO is defined as the total amount of time spent awake after falling asleep and before wake-up time as recorded in a sleep diary.
Difference of subjective number of awakenings (sNAW) between TS-142 and placebo in mean change from baseline | Baseline and Week 2
  sNAW is defined as the total number of awaking after falling asleep and before getting out of bed as recored in a sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No